CLINICAL TRIAL: NCT06958679
Title: A Phase I Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile, Immunogenicity, and Preliminary Anti-tumor Activity of SYS6005 in Patients With Advanced Malignant Tumor
Brief Title: Evaluation of SYS6005 in Patients With Advanced Malignant Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SYS6005-001
Record Dates: First submitted 2025-04-21; First posted 2025-05-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: B-cell Malignancies; Solid Tumors

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm, dose-escalation study using Bayesian Optimal Interval (BOIN) design. Seven dose levels will be tested. Dose-limiting toxicities (DLTs) will be assessed in Cycle 1 (21 days). The Safety Monitoring Committee (SMC) will review data to guide escalation. Pharmacokinetic analysis will use non-compartmental modeling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation and Dose expansion (Experimental): Participants will receive escalating doses of SYS6005 intravenously (IV) on Day 1 of each 21-day cycle in dose escalation phase and will receive selected doses of SYS6005 intravenously (IV) on Day 1 of each 21-day cycle in dose expansion phase
  Interventions: Drug: SYS6005

INTERVENTIONS:
Drug: SYS6005 — SYS6005 administered via IV infusion on , Day 1 of each 21-day cycle

SUMMARY:
This Phase I, open-label, multicenter study evaluates the safety, tolerability, pharmacokinetics, and preliminary efficacy of SYS6005 in advanced malignancies, comprising dose-escalation and expansion phases. The escalation phase employs a BOIN design with accelerated titration across seven dose levels, featuring a 21-day DLT observation period in Cycle 1, with dose adjustments guided by a Safety Monitoring Committee. In the expansion phase, one or more dosing regimens and tumor types will be selected, and participants will receive SYS6005 R2PD for further exploration and validation. Treatment continues until disease progression, unacceptable toxicity, or other discontinuation criteria. Safety monitoring includes AEs, labs, and ECOG PS, while efficacy is assessed via imaging. PK and immunogenicity samples are collected, and survival is tracked quarterly until death or study end. The study aims to determine the maximum tolerance dose (MTD)/recommended phase 2 dose (RP2D) and characterize SYS6005's clinical profile.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are voluntarily enrolled in this study and sign the informed consent form (ICF);
2. Age ≥ 18 years old, male or female;
3. Patients with advanced malignant tumors confirmed by cytology or histology, who have failed standard therapy or are intolerant to standard therapy and require systemic treatment： Solid tumor: Pathologically confirmed, unresectable advanced solid tumor with disease progression on or after at least 1 line of prior systemic therapy. Preferred tumor types include breast, lung, gynecologic, prostate, skin, adrenal, testicular, colon, bladder, pancreatic, gastric, kidney, cholangiocarcinoma, and esophageal cancers.

   B-cell malignancies: Pathologically confirmed Hodgkin and non-Hodgkin B-cell lymphoma as defined per 2016 WHO classification, with disease progression on or after at least 2 lines of prior systemic therapy. Preferred tumor types include cHL, DLBCL, MCL, FL, MZL, RTL, CLL/SLL;
4. Patients with at least one evaluable lesion as defined per RECIST v1.1 for solid tumor or 2014 Lugano Classification Criteria for lymphoma, respectively;
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0-2;
6. Expected survival ≥ 3 months;
7. Participants must have adequate organ function and have not received transfusion, erythropoietin, granulocyte colony-stimulating factor, or other medical supportive treatments within 14 days prior to examination
8. For participants enrolled in the dose-expansion phase, tumor tissue must be confirmed as ROR1-positive by the central laboratory during screening in order to be eligible for enrollment.
9. Male and female participants of childbearing potential must agree to use effective contraception from the time of signing the ICF until at least 6 months after the last dose of the investigational product; female participants of childbearing potential must have a negative pregnancy test result within 7 days prior to the first administration of the investigational product;
10. Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

1. Participants who have participated in other studies involving ROR1-targeted therapies prior to enrollment in this study, or have previously received ADC treatments containing MMAE payloads;
2. Participants with known central nervous system (CNS) lymphoma or CNS metastases from solid tumors that are symptomatic, untreated, or require treatment. Except for participants with metastases to CNS that have been completely resected and/or have stabilized or improved after radiotherapy, provided that imaging examinations prior to screening show stable disease for at least 4 weeks, and there is no evidence of brain oedema and no requirement for corticosteroids or anticonvulsant drugs;
3. Participants deemed suitable for CAR-T therapy or hematopoietic stem cell transplant (HSCT) by the investigator. Participants who have received an allogeneic haematopoietic stem cell transplant within 6 months prior to the first administration of the investigational product, have received an autologous haematopoietic stem cell transplant within 100 days prior to the first administration of the investigational product, or have received CAR-T cell therapy within 3 months prior to the first administration of the investigational product. Participants with active graft versus host disease;
4. Participants have a history of a second malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast or cancers that have been treated with no expectation of recurrence
5. Participants have a diagnosis of immunodeficiency, or has an active autoimmune disease or other conditions that require systemic steroid therapy For solid tumor: > 10 mg daily prednisone equivalents within 14 days prior to the administration of the first dose of SYS6005; For lymphoma: > 20 mg daily prednisone equivalents within 28 days prior to the administration of the first dose of SYS6005; The use of short-course systemic corticosteroids (≤ 7 days) is permitted, with a wash-out period of 1 week prior to the administration of the first dose of SYS6005
6. Participants with peripheral oedema, pericardial effusion, pleural effusion, or ascites that require medical intervention or limit daily life activities;
7. Participants with records of cerebrovascular events, angina unstable, myocardial infarction, or a history of NYHA Class III-IV cardiac symptoms within 6 months before the first administration of the investigational product, or a QTcF > 450 ms recorded in three repeated ECG examinations during screening;
8. Participants with any active infection requiring systemic treatment within 2 weeks prior to the first dose of investigational product;
9. Participants who have used strong inhibitors or inducers of CYP3A4 within 7 days prior to the first dose of the investigational product, or are expected to require the use of strong inhibitors or inducers of CYP3A4 during the study treatment;
10. Participants with the severity of any toxicities from prior treatments or surgery (excluding ≤ Grade 2 alopecia, endocrine disorders manageable with hormone replacement therapy, or other toxicities that the investigator considers do not pose a safety risk to the patient) has not returned to baseline or ≤ Grade 1 per NCI-CTCAE Version 5.0;
11. Participants with ≥ grade 2 peripheral neuropathy at baseline;
12. Participants who have received major surgery, radical radiotherapy, antibody-based targeted therapy, or immunotherapy within 28 days prior to the first administration of the investigational product, or who have received palliative radiation, chemotherapy, or small molecule targeted therapy within 14 days prior to the study treatment. Participants who have used anti-tumor Chinese herbal preparations or Chinese patent medicines within 14 days prior to the first administration of the investigational product;
13. Participants with history of immunodeficiency or positive human immunodeficiency virus (HIV) antibody test during screening;
14. Participants with active hepatitis B or hepatitis C, where active hepatitis B is defined as HBsAg positive and HBV DNA > 2000 IU/ml; active hepatitis C is defined as HCV antibody positive and HCV RNA > ULN;
15. Participants who have received a live vaccine within 28 days prior to the first dose of investigational product;
16. Participants with history of hypersensitivity or atopic reactions to excipients of the investigational product or any monoclonal antibodies;
17. Women who are pregnant or breastfeeding;
18. Other situations that may interfere with the participant's participation in the study program or are not in the participant's best interest or affect the study results include: history of mental illness, addiction or drug abuse, any other clinically significant illness or condition, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose limiting toxicities (for dose escalation part) | each cycle is 21 days
  A DLT is defined as a protocol pre-specified treatment-emergent adverse event (TEAE) that occurs in Cycle 1 of SYS6005 therapy and is considered drug-related.
Recommended Phase 2 Dose(RP2D) of SYS6005 (for dose escalation part) | About up to 6 months
  The selection of RP2D will be based on consideration of overall safety information together with available pharmacokinetic, pharmacodynamic, and efficacy data. The RP2D may be the MTD or may be a lower dose within the tolerable dose range.
Incidence and severity of adverse events (for both dose escalation and expansion part) | About up to 12 months
Overall response (for dose expansion part) | About up to 12 months
Complete remission (for dose expansion part) | About up to 12 months

SECONDARY OUTCOMES:
Pharmacokinetic (P K) profiles of SYS6005 including AUClast, AUCinf, Cmax, Tmax, t1/2, and CL, etc. | About up to 12 months
Immunogenicity of SYS6005： incidence and titer of ADAs, and incidence of neutralizing antibodies (Nabs) (if applicable) | About up to 12 months
Area Under the Concentration-Time Curve from Time Zero to the Last Quantifiable Concentration (AUClast) of SYS6005 | Cycle 1: Pre-dose, end of infusion (0,4,12,24,48,96,168,240,336 hours post); Cycle 2: Pre-dose, 0 hour post; Cycle 3: Pre-dose, end of infusion (0,4,12,24,48,96,168,240,336 hours post); Cycle 4: Pre-dose, 0 hour post
  AUClast reflects total drug exposure from administration to the last measurable concentration, calculated using the linear trapezoidal method.
Area Under the Concentration-Time Curve from Time Zero Extrapolated to Infinity (AUCinf) of SYS6005 | Cycle 1: Pre-dose, end of infusion (0,4,12,24,48,96,168,240,336 hours post); Cycle 2: Pre-dose, 0 hour post; Cycle 3: Pre-dose, end of infusion (0,4,12,24,48,96,168,240,336 hours post); Cycle 4: Pre-dose, 0 hour post
  AUCinf estimates total exposure by extrapolating AUClast using the terminal elimination rate (λz)
Maximum Observed Plasma Concentration (Cmax) of SYS6005 | Cycle 1: Pre-dose, end of infusion (0,4,12,24,48,96,168,240,336 hours post); Cycle 2: Pre-dose, 0 hour post; Cycle 3: Pre-dose, end of infusion (0,4,12,24,48,96,168,240,336 hours post); Cycle 4: Pre-dose, 0 hour post
  Peak plasma concentration, directly indicating the rate and extent of absorption
Time to Reach Maximum Plasma Concentration (Tmax) of SYS6005 | Cycle 1: Pre-dose, end of infusion (0,4,12,24,48,96,168,240,336 hours post); Cycle 2: Pre-dose, 0 hour post; Cycle 3: Pre-dose, end of infusion (0,4,12,24,48,96,168,240,336 hours post); Cycle 4: Pre-dose, 0 hour post
  Time point at which Cmax occurs, reflecting absorption kinetics.
Terminal Elimination Half-Life (t1/2) of SYS6005 | Cycle 1: Pre-dose, end of infusion (0,4,12,24,48,96,168,240,336 hours post); Cycle 2: Pre-dose, 0 hour post; Cycle 3: Pre-dose, end of infusion (0,4,12,24,48,96,168,240,336 hours post); Cycle 4: Pre-dose, 0 hour post
  Time for plasma concentration to reduce by 50% in the elimination phase, calculated as ln(2)/λz
Systemic Clearance (CL) of SYS6005 | Cycle 1: Pre-dose, end of infusion (0,4,12,24,48,96,168,240,336 hours post); Cycle 2: Pre-dose, 0 hour post; Cycle 3: Pre-dose, end of infusion (0,4,12,24,48,96,168,240,336 hours post); Cycle 4: Pre-dose, 0 hour post
  Volume of plasma cleared of drug per unit time (CL = Dose/AUCinf for IV administration).
Incidence of Anti-Drug Antibodies (ADAs) Against SYS6005 | Pre-dose on Day 1 of Cycles 1, 2, 3, 4; Pre-dose on Cycle 6; Pre-dose every 4 cycles thereafter (e.g., Cycle 10, 14, 18…); 30 days after last dose (follow-up).
  Proportion of subjects who develop detectable ADAs at any time during the study, expressed as a percentage.
Titer of Anti-Drug Antibodies (ADAs) Against SYS6005 | Pre-dose on Day 1 of Cycles 1, 2, 3, 4; Pre-dose on Cycle 6; Pre-dose every 4 cycles thereafter (e.g., Cycle 10, 14, 18…); 30 days after last dose (follow-up).
  Magnitude of ADA response (e.g., reported as geometric mean titer or median titer in ADA-positive subjects).
Incidence of Neutralizing Antibodies (NAbs) Against SYS6005 (if applicable) | Pre-dose on Day 1 of Cycles 1, 2, 3, 4; Pre-dose on Cycle 6; Pre-dose every 4 cycles thereafter (e.g., Cycle 10, 14, 18…); 30 days after last dose (follow-up).
  Proportion of subjects with NAbs capable of inhibiting SYS6005's pharmacological activity in a cell-based or competitive ligand-binding assay.

CONTACTS AND LOCATIONS:
Overall Officials: Qiu Lugui, Ph.D, Principal Investigator — Institute of hematology & blood disease hospital, Chinese academy of medical sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, China